CLINICAL TRIAL: NCT04989634
Title: Effects of Dietary and Weight Management on Pregnancy Outcomes in Mobile Medical Platform
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Capital Medical University (Other)
Responsible Party: Principal Investigator, Guanghui Li, Associate Professor, Capital Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2019-KY-036-02
Record Dates: First submitted 2021-07-26; First posted 2021-08-04 (Actual); Last update posted 2021-08-04 (Actual); Status verified 2021-07

CONDITIONS: Gestational Diabetes Mellitus; Hypertensive Disorder of Pregnancy
MeSH Terms: conditions — Diabetes, Gestational; Toxemia | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- standard care (Active Comparator): In the early pregnancy ( 8-12 weeks of pregnancy ) , a group education on dietary weight management will be carried out according to the current medical system and the regulations of our hospital , followed by routine prenatal examination . According to the corresponding diagnosis and treatment guidelines, examinations and follow-up interventions will be carried out if the metabolic diseases are occurred during pregnancy.
  Interventions: Behavioral: Standard care
- dietary and weight management (Experimental): A randomized controlled trial in pregnant women will be initiated at 8-12 weeks of gestation util delivery. The intervention contents included health education , nutritional analysis and individualized dietary guidance combined with mobile medical treatment and face-to-face teaching during the early , middle and late pregnancy stages.
  Interventions: Behavioral: Intensive dietary and weight management

INTERVENTIONS:
Behavioral: Intensive dietary and weight management — health education , nutritional analysis and individualized dietary guidance
  Arms: dietary and weight management
Behavioral: Standard care — Standard prenatal education on diet, nutrition and physical activity
  Arms: standard care

SUMMARY:
With the opening up of the two-child policy , the composition of pregnant women in China has changed significantly . The proportion of high-risk pregnant women in the elderly has increased significantly , and the risk of adverse pregnancy outcomes has also increased . Among them , gestational diabetes mellitus ( GDM ) is the most common complication during pregnancy . The incidence of GDM in China is as high as 18 % due to the economic growth , lifestyle changes and dietary habits . GDM not only threatens perinatal maternal and child health , but also increases the risk of offspring insulin resistance , obesity and metabolic diseases in adulthood . But it is still lack of experience on intervening and managing them effectively. Therefore , on the basis of previous studies , this study intends to explore the effects of intensive diet and exercise intervention by obstetricians and nutritionists on pregnancy weight gain , pregnancy outcome , glucose and lipid metabolism and postpartum weight retention under the mobile medical platform through a large sample cluster intervention test in the real world. In order to supervise and improve the compliance of the intervention subjects and realize the ultimate change of their behaviors, this study intends to use the APP software, the mobile medical technology, to monitor and evaluate diet , exercise and weight. Through the above research , it aims to improve the current management schemes of diet and weight during pregnancy , not only helps to optimize and improve the quality of perinatal health care , but also prevents the adult chronic diseases from the fetal period. This research has important theoretical and practical value .

DETAILED DESCRIPTION:
This is a cluster intervention study. A randomized controlled trial in pregnant women will be initiated at 8-12 weeks of gestation util delivery. Pregnant women who received routine antenatal examination in Beijing Obstetrics and Gynecology Hospital will be divided into two groups . One group contained 1000 cases as the control group , and the other group contained 1000 cases as a whole . The intervention contents included health education , nutritional analysis and individualized dietary guidance combined with mobile medical treatment and face-to-face teaching during the early , middle and late pregnancy stages. The primary outcome will be the incidence of GDM and the secondary outcome will be the incidence of hypertensive disorders of pregnancy , cesarean section , premature delivery , macrosomia, large for gestational age and so on.

ELIGIBILITY:
Inclusion Criteria:

* Regular check-ups in our hospital
* 18-44 years old
* 8-12 gestational weeks

Exclusion Criteria:

* Patients with incomplete medical records

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 2000 (Estimated)
Dates: Start 2019-07-01 (Actual); Primary Completion 2022-01-31 (Estimated); Study Completion 2022-01-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of gestational diabetes mellitus | From enrollment to 24-28 weeks of gestation

SECONDARY OUTCOMES:
Incidence of gestational hypertension | From date of randomization until the date of delivery, assessed up to 9 months
Incidence of cesarean section | From date of randomization until the date of delivery, assessed up to 9 months
Incidence of premature birth | From date of randomization until the date of delivery, assessed up to 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Guanghui Li, MD, PhD, Principal Investigator — Beijing Obstetrics and Gynecology Hospital
Locations (1):
- Beijing Obstetrics and Gynecology Hospital,Capital Medical University, Beijing, China